CLINICAL TRIAL: NCT01945645
Title: Ready to Act. A Health Education Programme for People With Screen-detected Hyperglycaemia
Brief Title: Ready to Act - Health Education in People With Hyperglycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Ready to Act; 20000183 (Other: Ethical approval)
Record Dates: First submitted 2013-09-14; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus; Behavior
Keywords: Prevention; Screening; Type 2 diabetes; Action Competence; Family practice; Health Services Research
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The Ready to Act programme aimed to promote health-related action competence including motivation, informed decision-making, action experience and social involvement The intervention was delivered across a number of primary care settings including the GP office, health centre and pharmacy. The programme consisted of two individual counselling interviews and eight group sessions, which totalled 18 hours within a three month period.
  Interventions: Behavioral: Ready to act

INTERVENTIONS:
Behavioral: Ready to act — The Ready to Act programme aimed to promote health-related action competence including motivation, informed decision-making, action experience and social involvement The intervention was delivered across a number of primary care settings including the GP office, health centre and pharmacy. The programme consisted of two individual counselling interviews and eight group sessions, which totalled 18 hours within a three month period.

SUMMARY:
A pre-randomized study in primary health care was designed to investigate health education in a subpopulation extracted from general practitioners (GPs) in one Danish county in the treatment arm of the ADDITION (Anglo-Danish-Dutch Study of Intensive Treatment in People with Screen-Detected Diabetes in Primary Care) study, DK. The overall objective of the 'Ready to Act' health education programme was to support the participants' competences in daily life and act appropriately with respect to their dysglycaemic condition. The achievement of action competence involved four learning objectives: intrinsic motivation, informed decision-making, action experience and social involvement. The programme was delivered in primary care settings (health centre or GP surgeries) by nurses, dieticians, physiotherapists and GPs.

ELIGIBILITY:
Inclusion Criteria:

* age 40-69 years at the time of screening and diagnosed with screen-detected T2D, IGT or IFG (according to WHO criteria).

Exclusion Criteria:

* women who were pregnant or lactating, those with a psychotic illness or an illness with a prognosis of less than one year.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Modelled cardiovascular disease risk | 3 years after intervention, dec 2010
  The risk is measured by a SCORE model uses information on age, sex, smoking status, total cholesterol and systolic blood pressure. It provides an estimate of ten-year fatal cardiovascular disease risk

SECONDARY OUTCOMES:
Glycated hemoglobin | 3 years after intervention, dec 2010
  Glycated hemoglobin (HbA1c)is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time
se-cholesterol | 3 years after intervention, dec 2010
  Serum cholesterol is the total amount of cholesterol found in the blood.
Patient Activation | One year and three year (2006, 2007, 2010)
  The Patient Activation Measure (PAM-13) is a composite measure of perceived skills, self-efficacy and knowledge.
Blood pressure | 3 years after intervention, dec 2010
  Systolic and diastolic blood pressure were measured
Physical activity | 3 years after intervention, dec 2010
  Physical activity was measured using the International Physical Activity questionnaire (IPAQ-short form)
Smoking | 3 years after intervention, 2010
  Smoking status was assessed by standard questions.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Terkildsen Maindal, MPH, PhD, Principal Investigator — Aarhus university, Department of Public health
Locations (1):
- Department of Public health, Aarhus, Denmark